CLINICAL TRIAL: NCT06337279
Title: The Clinical Value of Systemic Oxidative Stress Score in Predicting Long-term Survival and Recurrence Risk in Gastric Cancer: A Multicenter Real-world Cohort Study
Brief Title: Systemic Oxidative Stress Score as a Predictor of Gastric Cancer Survival and Recurrence Risk
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Collaborators: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: FMUUH-0322
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
Keywords: Oxidative stress; Gastric cancer; Recurrence; Disease-free survival; Systemic Oxidative Stress Score
MeSH Terms: conditions — Stomach Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Systemic Oxidative Stress Score (SOSS) , a comprehensive score reflecting the oxidative stress conditions in the microenvironment, can independently and effectively predict tumor burden and long-term prognosis in GC patients. Nomograms based on SOSS provide a potential and promising model for risk stratification and guiding the implementation of treatment decisions.

DETAILED DESCRIPTION:
We retrospectively analyzed the clinical data of gastric cancer patients who underwent radical gastrectomy in three hospitals from January 2009 to June 2020. The data from one hospital were randomly divided into a training cohort and an internal validation cohort in a 7:3 ratio, while the data from the other two centers were used as an external validation cohort. In the training cohort, COX proportional risk models were employed to identify key indicators of SOSS and independent prognostic factors influencing patients' OS and DFS. Subsequently, based on the results of the multifactor COX analysis, two predictive models for OS and DFS were developed. The predictive efficacy, calibration, and clinical utility of the models were evaluated using ROC curves, calibration curves, and decision curves in the internal and external validation cohorts, respectively. Both models demonstrated good discriminative ability between postoperative survival and recurrence risk, outperforming TNM staging in terms of predictive accuracy.

ELIGIBILITY:
Inclusion Criteria:

1) gastroscopic histopathological diagnosis of gastric adenocarcinoma; 2) radical gastrectomy for GC; 3) preoperative examination of oxidative indicators including Fbg, CHOL, ALB, TBIL, DBIL, and CR within seven days before surgery; and 4) the tumor did not invade neighboring organs or had no distant metastasis.

Exclusion Criteria:

1) gastroscopic histopathological diagnosis of non-adenocarcinoma, 2) gastric stump cancer, 3) neoadjuvant chemotherapy, 4) other malignant diseases besides GC, 5) incomplete medical records, and 6) patients with GC lost to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a multicenter, retrospective cohort investigation involving GC patients who underwent radical gastrectomy at the Fujian Medical University Union Hospital (FMUUH), the First Affiliated Hospital of Gannan Medical University (FAHGMU) and Quzhou Affiliated Hospital of Wenzhou Medical University (QAHWMU) between January 2009 and June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 3820 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
5-year OS | 5 years or 60 months
  Overall survival, death, survival with tumor, deletion.
5-year DFS | 5 years or 60 months
  Disease-free survival, death,recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Prof., Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China